CLINICAL TRIAL: NCT05559411
Title: A Prospective Non-interventional Multicenter Cohort Study to Evaluate Different Imaging-guided Methods for Localization of Non-palpable Malignant Breast Lesions
Brief Title: MEthods for LOcalization of Different Types of Breast Lesions
Acronym: MELODY
Status: Recruiting | Type: Observational
Sponsor: European Breast Cancer Research Association of Surgical Trialists (Network)
Collaborators: iBRA-NET (Unknown)
Responsible Party: Sponsor
Other Study IDs: EUBREAST-4
Record Dates: First submitted 2022-09-18; First posted 2022-09-29 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; non-palpable breast lesion; localization technique; localization device; intraoperative ultrasound; patient-reported outcome
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- Wire-guided Localization
- Intraoperative Ultrasound
- Magnetic Localization
- Radar Reflector Localization
- Radiofrequency Localization
- Radioactive Localization
- Ink Localization
- Luminomark Localization

SUMMARY:
In the last decades, the proportion of breast cancer (BC) patients receiving breast-conserving surgery has increased steadily, reaching 70-80% in developed countries. Since positive resection margins are strongly associated with local recurrence risk, the goal of breast surgery is the complete tumor removal and most national and international guidelines recommend re-operation, either in form of re-excision or mastectomy, until clear margins have been reached. Re-operation rates vary widely, with population-based studies reporting a range of 15-35%, and the necessity for a second surgery can lead to increased patient anxiety, a delay in start of adjuvant treatment, worse cosmetic outcome and increased complication rates and costs. Therefore, re-operation rate has been included as a quality indicator in several countries.

Several imaging-guided techniques have been developed to guide removal of non-palpable breast lesions, the oldest one being preoperative wire placement under ultrasound or mammographic guidance, usually followed by radiography or ultrasound of removed tissue. Newer techniques, such as intraoperative ultrasound (IOUS), radioguided occult lesion localization (ROLL), radioactive seed localization (RSL), radar reflector-localization (RRL), magnetic seed localization (MSL), and radiofrequency identification (RFID) tags have been introduced as an alternative to wire-guided localization (WGL).

To date, comparative data on the rates of successful lesion removal, negative margins, re-operation rate and patient's comfort depending on the localization technique used are limited. Further, since some of these studies were funded by the manufacturer of the marker examined, a potential bias cannot be excluded. In the vast majority of the available studies, the patient's perspective with regard to discomfort and pain level has not been evaluated.

The aim of the proposed study is to comparatively evaluate different imaging-guided localization methods used for surgical removal of malignant breast lesions with regard to oncological safety and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Malignant breast lesion requiring breast-conserving surgery and imaging-guided localization (either DCIS or invasive breast cancer; multiple or bilateral lesions and the use of neoadjuvant chemotherapy are allowed)
* Planned surgical removal of the lesion using one or more of the following imaging-guided localization techniques:

  * Wire-guided localization
  * Intraoperative ultrasound
  * Magnetic localization
  * Radioactive seed localization
  * Radioguided Occult Lesion Localization (ROLL)
  * Radar localization
  * Radiofrequency identification (RFID) tag localization
  * Ink/carbon localization
* Female / male patients ≥ 18 years old

Exclusion Criteria:

* Patients not suitable for surgical treatment
* Patients requiring mastectomy as first surgery
* Surgical removal without imaging-guided localization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male patients with invasive breast cancer or DCIS scheduled for breast-conserving surgery with an imaging-guided localization
Sampling Method: Probability Sample
Enrollment: 7416 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of intended target lesion and/or marker removal, independent of margin status on final histopathology (number of study participants with intended target lesion and/or marker removal, divided by the number of all study participants) | 2 years
Negative resection margin rates (defined as lesion removal with no invasive or non-invasive carcinoma on ink) at first surgery | 2 years
  Number of study participants with a negative resection margin, divided by the number of all study participants

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Schleswig-Holstein Campus Lübeck, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.eubreast.com/index.php?Trials/MELODY